CLINICAL TRIAL: NCT00942370
Title: Comparison of Electromyographic With Mechanomyographic Signals of Rectus Abdominis
Brief Title: Electromyographic (EMG) and Mechanomyographic (MMG) Comparison
Acronym: EMG-MMG
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: DCIC 0904
Record Dates: First submitted 2009-07-02; First posted 2009-07-20 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Stress Urinary Incontinence
Keywords: mechanography; electromyography; effort cough
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- accelerometric device
  Interventions: Device: non invasive mechanomyographic device based on a 3 axes accelerometer

INTERVENTIONS:
Device: non invasive mechanomyographic device based on a 3 axes accelerometer — This biomedical research consists specifically in the simultaneous acquisition of:
  * EMG and MMG Signals of rectus abdominis of the abdomen,
  * Respiratory flow,
  * An electrocardiogram (ECG).
  These acquisitions will be conducted on 16 healthy volunteers according to a standardized protocol, at rest and during voluntary cough and various physical exercises often resulting in urinary leakage in the incontinent person.

SUMMARY:
The purpose of this study is to assess the delay between the detection (by mechanomyography-MMG) of rectus abdominis contraction and the detection of cough in cough effort.

ELIGIBILITY:
Inclusion Criteria:

* More or equal than 18 years old
* Patient affiliated to social security or similarly regime
* Healthy volunteer
* BMI less than 30

Exclusion Criteria:

* Pregnant women and lactating mothers
* Ward of court or under guardianship
* Adult unable to express their consent or person under legal protection
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Delay between the detection by mechanomyography (MMG) of rectus abdominis contraction and the detection of cough in cough effort | 2 hours

SECONDARY OUTCOMES:
Lower and upper spectral band frequencies values for which the majority of the MMG signal is present, thresholds for detection of rectus abdominis contraction by mechanical myography | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Moreau-Gaudry, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Clinical Investigation Center - INSERM - University Hospital of Grenoble, Grenoble, France

REFERENCES:
- See also: Related Info — http://www.cic-it-grenoble.fr/